CLINICAL TRIAL: NCT00072293
Title: A Randomized Trial Of Axillary Dissection Versus No Axillary Dissection For Patients With Clinically Node Negative Breast Cancer And Micrometastases In The Sentinel Node
Brief Title: Surgical Resection With or Without Axillary Lymph Node Dissection in Treating Women With Node-Negative Breast Cancer and Sentinel Lymph Node Micrometastases
Acronym: 23-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000339581; IBCSG 23-01 (Other: IBCSG)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Axillary Dissection (Active Comparator): Patients undergo surgical resection of the primary tumor with axillary lymph node dissection following sentinel lymph node assessment.
  Interventions: Procedure: Axillary lymph node dissection
- No Axillary Dissection (Experimental): Patients undergo surgical resection of the primary tumor with no axillary lymph node dissection following sentinel lymph node assessment.
  Interventions: Procedure: No axillary lymph node dissection

INTERVENTIONS:
Procedure: Axillary lymph node dissection — Axillary lymph node dissection
  Arms: Axillary Dissection
Procedure: No axillary lymph node dissection — Therapeutic conventional surgery
  Arms: No Axillary Dissection

SUMMARY:
RATIONALE: Surgery to remove lymph nodes in the armpit in patients with sentinel lymph node micrometastases may remove cancer cells that have spread from tumors in the breast. It is not yet known whether surgery to remove the primary tumor is more effective with or without axillary lymph node dissection.

PURPOSE: This randomized phase III trial is studying surgery and axillary lymph node dissection to see how well they work compared to surgery alone in treating women with node-negative breast cancer and sentinel lymph node micrometastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival of women with clinically node-negative breast cancer with sentinel lymph node micrometastases treated with surgical resection with or without axillary dissection.
* Compare overall survival of patients treated with these regimens.
* Assess sites of recurrence, particularly reappearance of disease in the undissected axilla.
* Assess long-term surgical complications in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, menopausal status (pre- vs postmenopausal), and preoperative sentinel node biopsy (yes vs no). Patients are followed every 4 months for 1 year, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical, mammographic, ultrasonographic, or pathologic diagnosis of unicentric and unifocal breast carcinoma
* Largest tumor lesion ≤ 5 cm
* Palpable or nonpalpable breast lesion

  * Preoperative radioactive occult lesion localization, hook wire, or other method of localization required for nonpalpable lesions
* Prior (preoperative) or planned (intraoperative) sentinel node biopsy required

  * At least 1 micrometastatic (i.e., no greater than 2 mm) sentinel lymph node with no extracapsular extension
* No clinical evidence of distant metastases

  * No suspicious manifestation of metastases that cannot be ruled out by x-ray, MRI, or CT scan, including the following:

    * Skeletal pain of unknown cause
    * Elevated alkaline phosphatase
    * Bone scan showing hot spots
* No palpable axillary lymph node(s)
* No Paget's disease without invasive cancer
* Hormone receptor status:

  * Estrogen receptor and progesterone receptor known

PATIENT CHARACTERISTICS:

Age

* Any age

Sex

* Female

Menopausal status

* Any status

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* See Disease Characteristics

Renal

* Not specified

Other

* Not pregnant or nursing
* No other prior or concurrent malignancy except the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated carcinoma in situ of the cervix
  * Adequately treated in situ melanoma
  * Contralateral or ipsilateral carcinoma in situ of the breast
* No psychiatric, addictive, or other disorder that may compromise ability to give informed consent
* Geographically accessible for follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No prior systemic therapy for breast cancer
* More than 1 year since prior chemopreventive agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 931 (Actual)
Dates: Start 2001-12; Primary Completion 2012-09 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viviana E. Galimberti, Study Chair — European Institute of Oncology; Umberto Veronesi, MD, Prof., Study Chair — European Institute of Oncology
Locations (31):
- Australia (10):
  - Lismore Base Hospital, Lismore, New South Wales
  - St Vincents Hospital, Lismore, New South Wales
  - Mater Hospital - North Sydney, North Sydney, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital Cancer Centre, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - St. John of God Hospital - Bunbury, Bunbury, Western Australia
- CHU Liege - Domaine Universitaire du Sart Tilman, Liège, Belgium
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Horsholm Sygenus, Hørsholm, Denmark
- Institut Gustave Roussy, Villejuif, France
- Italy (8):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedali Riuniti di Bergamo, Bergamo
  - University of Bologna Medical School, Bologna
  - Universita di Ferrara, Ferrara
  - Ospedale Alessandro Manzoni, Lecco
  - Istituto Scientifico H. San Raffaele, Milan
  - European Institute of Oncology, Milan
  - Fondazione Salvatore Maugeri, Pavia
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Waikato Hospital, Hamilton
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- Switzerland (5):
  - Kantonspital Aarau, Aarau
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen

REFERENCES:
- [Derived] Galimberti V, Cole BF, Viale G, Veronesi P, Vicini E, Intra M, Mazzarol G, Massarut S, Zgajnar J, Taffurelli M, Littlejohn D, Knauer M, Tondini C, Di Leo A, Colleoni M, Regan MM, Coates AS, Gelber RD, Goldhirsch A; International Breast Cancer Study Group Trial 23-01. Axillary dissection versus no axillary dissection in patients with breast cancer and sentinel-node micrometastases (IBCSG 23-01): 10-year follow-up of a randomised, controlled phase 3 trial. Lancet Oncol. 2018 Oct;19(10):1385-1393. doi: 10.1016/S1470-2045(18)30380-2. Epub 2018 Sep 5. PMID 30196031
- [Derived] Galimberti V, Cole BF, Zurrida S, Viale G, Luini A, Veronesi P, Baratella P, Chifu C, Sargenti M, Intra M, Gentilini O, Mastropasqua MG, Mazzarol G, Massarut S, Garbay JR, Zgajnar J, Galatius H, Recalcati A, Littlejohn D, Bamert M, Colleoni M, Price KN, Regan MM, Goldhirsch A, Coates AS, Gelber RD, Veronesi U; International Breast Cancer Study Group Trial 23-01 investigators. Axillary dissection versus no axillary dissection in patients with sentinel-node micrometastases (IBCSG 23-01): a phase 3 randomised controlled trial. Lancet Oncol. 2013 Apr;14(4):297-305. doi: 10.1016/S1470-2045(13)70035-4. Epub 2013 Mar 11. PMID 23491275
- See also: Abstract from paper published in Lancet Oncology, 2013 — http://www.ncbi.nlm.nih.gov/pubmed/23491275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual began April 1, 2001 and closed February 28, 2010, after 934 patients from 27 centers in Europe, South America and Australia were randomized.
Period: Overall Study
Arm/Group | Axillary Dissection | No Axillary Dissection
Started | 465 | 469
Completed | 464 | 467
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Axillary Dissection | No Axillary Dissection | Total
Number analyzed (Participants) | 464 | 467 | 931
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [28 to 81] | 54 [26 to 81] | 54 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 464 | 467 | 931
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 5-year Disease-Free Survival
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where disease-free survival is defined as the time from randomization to first evidence of invasive relapse at any site, second primary tumor (contralateral or non-breast) or death.
Time Frame: 5-year estimate reported after a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Axillary Dissection | No Axillary Dissection
Number analyzed (Participants) | 464 | 467
percentage of participants | 84.4 | 87.8
Statistical Analysis 1: Comparison: Axillary Dissection vs No Axillary Dissection; Test type: Non-Inferiority or Equivalence — As originally designed, target accrual was 1960 patients with analysis planned after 558 events. These targets were based on having 90% power to detect non-inferiority of no axillary dissection with a one-sided statistical signifi cance level of 10% (ie, α=0·10) under the assumption that 5-year disease-free survival with axillary dissection was 70% and defining non-inferiority as a hazard ratio (HR) of less than 1·25 (no axillary dissection relative to axillary dissection); p = 0.004, 1-sided non-inferiority test — Test for non-inferiority of no axillary dissection. Stratified logrank test compared groups. HR (no-AD vs AD) estimated from test statistic and variance as HR=exp([O-E]/V), compared to 1.25 in 1-sided test of non-inferiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.55 to 1.11] — Hazard Ratio is no axillary dissection/axillary dissection

2. Secondary Outcome: 5-year Overall Survival
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where overall survival is defined as the time from randomization to death of any cause.
Time Frame: 5-year estimate reported after a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Axillary Dissection | No Axillary Dissection
Number analyzed (Participants) | 464 | 467
percentage of participants | 97.6 | 97.5
Statistical Analysis 1: Comparison: Axillary Dissection vs No Axillary Dissection; Test type: Superiority or Other; p = 0.73, Log Rank; Hazard Ratio (HR) = 0.89, 90% CI 2-sided [0.52 to 1.54] — Hazard Ratio is no axillary dissection/axillary dissection

3. Secondary Outcome: Site of Recurrence
Description: Site of recurrence of breast cancer
Time Frame: Reported after a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Axillary Dissection | No Axillary Dissection
Number analyzed (Participants) | 464 | 467
participants
  Local recurrence | 10 | 8
  Regional recurrence | 1 | 5
  Contralateral breast cancer | 3 | 9
  Distant recurrence | 34 | 25
  Second (non-breast) primary | 20 | 6
  Death without cancer event | 1 | 2

ADVERSE EVENTS:
Time Frame: 5-years. Treating physician assessed and reported long-term surgical events (sensory neuropathy, lymphoedema and motor neuropathy) at every follow-up visit (every 4 months from date of randomization for the first year and every six months from years 2-5).
Description: Analysis population excludes 31 patients (17 in Axillary Dissection group/14 in No Axillary Dissection group) who did not receive the randomly-assigned treatment.
Arm/Group | Axillary Dissection | No Axillary Dissection
Serious Adverse Events (participants affected / at risk) | 1/447 | 0/453
Other Adverse Events (participants affected / at risk) | 178/447 | 83/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axillary Dissection (N=447) | No Axillary Dissection (N=453)
Post-operative infection (L.axilla) (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axillary Dissection (N=447) | No Axillary Dissection (N=453)
Sensory neuropathy (Nervous system disorders) | 82 | 55
Lymphedema (Vascular disorders) | 59 | 15
Motor neuropathy (Nervous system disorders) | 37 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No